CLINICAL TRIAL: NCT00247936
Title: Combined Thoracoscopic and Laparoscopic Esophagectomy vs. Hand-assisted Transhiatal Esophagectomy: A Prospective Trial.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Prior to recruitment, study terminated lack of recruitment interest.
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS 2003-3422
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinoma
Keywords: Adenocarcinoma, Esophagectomy
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Combined Thoracoscopic and Laparoscopic Esophagectomy
  Interventions: Procedure: Laparoscopic Esophagectomy
- 2 (Active Comparator): Hand-Assisted Transhiatal Esophagectomy
  Interventions: Procedure: Laparoscopic Esophagectomy

INTERVENTIONS:
Procedure: Laparoscopic Esophagectomy — Laparoscopic Esophagectomy
  Other Names: Laparoscopic Esophagectomy; Hand-Assisted Transhiatal Esophagectomy

SUMMARY:
Esophagectomy for benign or malignant disease of the esophagus can be performed using a transhiatal technique or Ivor Lewis technique (combined laparotomy with thoracotomy). These procedures can be associated with significant morbidity and mortality [1]. Advances in minimally invasive technology and surgical techniques have allowed us to explore the possibility of performing esophagectomy using minimally invasive surgical techniques.

Minimally invasive esophagectomy represents a new alternative to conventional open esophagectomy. It is a technically demanding operation requiring advanced laparoscopic surgical skills, appropriate instrumentation, and thorough knowledge of open esophagectomy. Multiple authors have reported the use of video-assisted thoracoscopy or laparoscopy to facilitate esophagectomy [2-6]. Most of these reports have utilized a standard laparotomy in combination with thoracoscopy to perform esophageal mobilization or laparoscopy with a mini-laparotomy to perform esophagectomy. DePaula was the first to report a large series of 48 patients undergoing laparoscopic transhiatal esophagectomy for benign (n=24) and malignant disease (n=24) [7]. In 2 patients, conversion to open surgery was required and 2 others required thoracoscopic assistance. Postoperative complications were low in the benign group but higher in the carcinoma group. The 30-day mortality rate was 16% in patients with carcinoma undergoing laparoscopic transhiatal esophagectomy. DePaula concluded that the patients who benefit most from this procedure are those with benign disease. Swanstrom recently reported nine cases of laparoscopic total esophagectomy [8]. There were no conversions to laparotomy. One patient required a right thoracoscopy with intrathoracic anastomosis due to poor viability of the gastric tube. The mean operative time was 6.5 hours with a mean hospital stay of 6.4 days. However, the advantages of minimally invasive esophagectomy have not been observed. The aim of this prospective trial is to evaluate the physiologic outcome, clinical outcome, and quality of life after combined thoracoscopic and laparoscopic esophagectomy vs. transhiatal esophagectomy.

DETAILED DESCRIPTION:
RATIONALE:

Open esophagectomy can be associated with significant morbidity. We hypothesize that laparoscopic esophagectomy is associated with reduced morbidity and a faster recovery.

HYPOTHESES:

1. Combined thoracoscopic and laparoscopic esophagectomy can be performed safely.
2. Combined thoracoscopic and laparoscopic esophagectomy is associated with reduced postoperative pain, decrease ICU and hospital stay, and reduced postoperative wound morbidity.
3. Combined thoracoscopic and laparoscopic esophagectomy is associated with similar long term survival as with the open approach for patients with esophageal malignancies.

OBJECTIVES AND SPECIFIC AIMS:

1. To compare short-term outcome such as operative time, operative and in-patient costs, operative complications, length of hospital stay, and postoperative complications between combined thoracoscopic/ laparoscopic esophagectomy and transhiatal esophagectomy.
2. To evaluate physiologic outcomes after minimally invasive esophagectomy vs. transhiatal esophagectomy.
3. To determine the long-term outcome, disease-free survival, survival and quality of life after minimally invasive esophagectomy compared to transhiatal esophagectomy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy proven esophageal malignancies
2. Patients with recalcitrant severe esophageal stricture
3. Karnofsky score >60
4. No previous treatment for any other cancer over the past 2 years (except for skin cancer)

Exclusion Criteria:

1. Malignant tracheoesophageal fistula or presence of tracheal involvement
2. Unacceptable operative risk
3. Tumor size greater than 12 centimeters.
4. Tumor involvement of the aorta or trachea.
5. Renal or liver insufficiency (Creatinine > 2.0, transaminase > fourfold)
6. WBCs <2,000, platelets <80,000
7. Presence of metastatic disease
8. Patients with previous esophageal resection
9. Minors and pregnant women are excluded. The chance of esophageal cancer presenting in anyone under 18 years of age is essentially null. Pregnant women are excluded because of safety for the fetus.

   * All physician, hospital, surgery, and laboratory costs will be billed to the subject and/or their insurance carrier as customary for they are considered standard of care procedures. All research-related procedures such as pulmonary function tests and study questionnaires conducted in this study will be paid for by the primary investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-05; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
short-term surgical outcome of minimally invasive esophagectomy vs. transhiatal esophagectomy | 30-day

SECONDARY OUTCOMES:
long-term surgical outcome of minimally invasive esophagectomy vs. transhiatal esophagectomy. | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Ninh T Nguyen, MD, Principal Investigator — University of California, Irvine